CLINICAL TRIAL: NCT00944151
Title: Continuous Transversus Abdominis Plane Nerve Block for Postoperative Analgesia: A Randomized, Triple-Masked, Placebo-Controlled Study
Brief Title: Continuous Transversus Abdominis Plane Nerve Block for Postoperative Analgesia
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: lack of enrollment
Sponsor: University of California, San Diego (Other)
Responsible Party: Vanessa Loland/Principal Investigator, University of California, San Diego, Department of Anesthesiology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAP Catheter
Record Dates: First submitted 2009-07-21; First posted 2009-07-23 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2009-07

CONDITIONS: Incisional Pain
Keywords: pain; UCSD; catheter; nerve block; hernia; post-surgery pain; abdominal pain; pelvic pain; Transversus abdominal plane; Hernia Repair; Transversus Abdominal Plane Block
MeSH Terms: conditions — Pain; Hernia; Abdominal Pain; Pelvic Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single injection with Saline infused TAP catheter (Placebo Comparator): Prior to surgery patient will receive single injection of 0.5% ropivacaine and a TAP catheter. Following surgery patient will be given normal saline in infusion pump, attached to catheter.
  Interventions: Procedure: TAP Catheter and Infusion of Study Solution
- Single injection with Ropivicaine infused TAP catheter (Active Comparator): Prior to surgery patient will receive single injection of 0.5% ropivacaine and a TAP catheter. Following surgery patient will be given 0.2% ropivicaine in infusion pump, attached to catheter
  Interventions: Procedure: TAP Catheter and Infusion of Study Solution

INTERVENTIONS:
Procedure: TAP Catheter and Infusion of Study Solution — Subject will be randomized to one of two groups: Saline infused TAP catheter following surgery for 0-2 days or ropivacaine infused TAP catheter following surgery for 0-2 days. All patients will be given a single injection of ropivacaine prior to surgery. Research staff will follow all patients for two days following surgery or while they have TAP catheter in.

SUMMARY:
Research study to determine if putting local anesthetic through one or two tiny tubes next to the nerves that go to the area the patients are having surgery on (abdomen or pelvis), will improve pain control following surgery. This study will also help determine if patients require fewer pain pills, experience fewer sleep disturbances, and are more satisfied with their postoperative pain control.

DETAILED DESCRIPTION:
Specific Aim: To determine if adding a continuous Transversus Abdominis Plane nerve block to a single-injection nerve block results in improved postoperative pain control.

Hypothesis 1: Adding a continuous Transversus Abdominis Plane nerve block to a single-injection nerve block results in lower average pain scores during movement the day following surgery.

Specific Aim2: To determine if adding a continuous Transversus Abdominis Plane nerve block to a single-injection nerve block results in decreased average pain scores, opioid use, sleep disturbances, and improved patient satisfaction.

Hypothesis 2: Adding a continuous Transversus Abdominis Plane nerve block to a single-injection nerve block results in decreased average pain scores, oral opioid consumption, sleep disturbances, and improved patient satisfaction the day following surgery.

ELIGIBILITY:
Inclusion Criteria:

* undergoing ambulatory inguinal and/or abdominal surgery amenable to a Transversus Abdominis Plane nerve block (unilateral or bilateral).
* expected postoperative pain to be at least moderate in severity the day following surgery
* age 18 years or older
* desires a regional anesthetic for postoperative analgesia
* is able to understand the possible perineural infusion-related complications, study protocol, and catheter/pump care
* has a caretaker through the first night after surgery
* has an ASA Physical Status Classification of 1-3

Exclusion Criteria:

* any contraindication for a continuous Transversus Abdominis Plane nerve block
* any physical, mental or medical conditions which, in the opinion of the investigators, may confound quantifying postoperative pain resulting from surgery.
* current chronic opioid or tramadol use
* history of alcohol or opioid abuse
* know allergy or other contraindication to the study medication
* pregnancy
* known hepatic or renal insufficiency/disease
* peripheral neuropathy of the surgical site
* morbid obesity
* inability to communicate with the investigators and hospital staff
* incarceration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-07; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
The primary outcome measurement will be the average pain with movement on postoperative day 1 as measured by 0-10 scale, where 0=no pain and 10=worst imaginable pain. | 1 day

SECONDARY OUTCOMES:
Pain with movement on second day following surgery, as measured by 0-10 scale (where 0=no pain and 10=worst imaginable pain). | 2 days
Total opioid consumption per day following surgery as measured by the number of opioid pills consumed per day. | Day 1 and 2 following surgery
Sleep disturbances, measured on days 1 and 2 following surgery, as asked by research staff during follow-up phone calls. | Days 1 and 2 following surgery
Patient satisfaction of pain control as measured on a 0-10 scale where 0=very unsatisfied and 10=very satisfied with pain control | Day 2 following surgery

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Loland, M.D., Principal Investigator — University of California, San Diego
Locations (1):
- UCSD Medical Center, San Diego, California, United States